CLINICAL TRIAL: NCT01028768
Title: Open Label Pharmacokinetic (PK) Study, Conducted at One Investigational Site in Germany, to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of Teduglutide Following Subcutaneous Administration of 10 mg Teduglutide and to Evaluate Safety and Tolerability of 10 mg Teduglutide
Brief Title: Pharmacokinetics of 10 mg Teduglutide in Subjects With Renal Impairment Compared to Healthy Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nycomed (Industry)
Collaborators: NPS Pharma (Industry)
Responsible Party: Head of Exploratory Clinical Development, Nycomed GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TE-1777-101-EC
Record Dates: First submitted 2009-12-03; First posted 2009-12-09 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2010-04

CONDITIONS: Renal Impairment
Keywords: Renal impairment; Renal impairment study
MeSH Terms: conditions — Renal Insufficiency | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teduglutide (Experimental)
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — 10 mg, one-time subcutaneous

SUMMARY:
To evaluate the effect of renal impairment on the pharmacokinetics (PK) of teduglutide following subcutaneous (SC) administration of 10 mg teduglutide.

Secondary objectives are to assess the safety and tolerability of 10 mg teduglutide. A further objective is the description of the PK of teduglutide following SC administration of 10 mg teduglutide in elderly (≥ 65 years) healthy subjects compared to non elderly healthy subjects.

DETAILED DESCRIPTION:
Pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate, severe and end stage renal failure and matched healthy controls.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of teduglutide | 24 hrs

SECONDARY OUTCOMES:
Safety and tolerability of 10 mg teduglutide (assessed by physical examination, vital signs, clinical laboratory, electrocardiogram [ECG] and adverse events [AE]) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nycomed GmbH, Konstanz, Germany